CLINICAL TRIAL: NCT06929897
Title: Comparison of Pulmonary Vein Isolation Alone Versus Pulmonary Vein Isolation With Posterior Wall Isolation for Pulse-Field Ablation in Persistent Atrial Fibrillation: A Prospective Randomized Controlled Trial
Brief Title: PVI Alone vs PVI With Posterior Wall Isolation for Pulse-Field Ablation in Persistent AF
Acronym: POBI-PFA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Collaborators: Ewha Womans University Seoul Hospital (Other); Korea University Anam Hospital (Other); Ajou University School of Medicine (Other); Seoul National University Bundang Hospital (Other); Kangbuk Samsung Hospital (Other); Hanyang University Seoul Hospital (Other); Asan Medical Center (Other); Wonkwang University Hospital (Other); Korea University Guro Hospital (Other); Severance Hospital (Other); Eunpyeong St. Mary's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POBI-PFA
Record Dates: First submitted 2025-03-13; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation (AF)
Keywords: pulsed field ablation; catheter ablation; posterior wall isolation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Pulmonary vein isolation (PVI) is performed using pulsed-field ablation. Afterward, electrical cardioversion is performed to restore normal sinus rhythm. Patients who successfully convert to sinus rhythm are then randomly assigned to either the PVI-only group or the PVI with additional left atrial posterior wall isolation group.
  1. Patients requiring catheter ablation for persistent atrial fibrillation (AF).
  2. AF ablation is performed while maintaining anticoagulation therapy.
  3. Pulmonary vein isolation (PVI) is performed as the primary procedure.
  4. After PVI, direct current (DC) cardioversion is performed to restore normal sinus rhythm. If the patient converts to sinus rhythm, they are randomly assigned to either the PVI-only group or the additional left atrial posterior wall ablation group.
  5. Patients who fail to convert to sinus rhythm after DC cardioversion are excluded from randomization.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Additional Left Atrial Posterior Wall Ablation Group (Active Comparator): After pulmonary vein isolation, electrical isolation of the left atrial posterior wall is performed using a pulsed-field ablation catheter with EGM-guided ablation.
  Interventions: Procedure: Pulmonary Vein Isolation; Procedure: Additional Left Atrial Posterior Wall Ablation
- Pulmonary Vein Isolation (PVI) only Group (Placebo Comparator): Electrical isolation of all four pulmonary veins is performed using a pulsed-field ablation catheter.
  Interventions: Procedure: Pulmonary Vein Isolation; Procedure: Non-PV trigger test

INTERVENTIONS:
Procedure: Pulmonary Vein Isolation — 1. Pulmonary vein isolation (PVI) is performed as the primary procedure.
  2. After PVI, direct current (DC) cardioversion is performed to restore normal sinus rhythm. If the patient converts to sinus rhythm, they are randomly assigned to either the PVI-only group or the additional left atrial posterior wall ablation group.
  3. Patients who fail to convert to sinus rhythm after DC cardioversion are excluded from randomization.
  Other Names: PVI
Procedure: Additional Left Atrial Posterior Wall Ablation — 1. Additional left atrial posterior wall ablation is performed.
  2. Complete electrical isolation of the entire left atrial posterior wall is confirmed (posterior box lesion isolation must be achieved).
  3. Post-procedural rhythm monitoring follows the study protocol.
  Other Names: Posterior box isolation
  Arms: Additional Left Atrial Posterior Wall Ablation Group
Procedure: Non-PV trigger test — 1. If atrial fibrillation triggers are identified with isoproterenol infusion, additional focal ablation is performed.
  2. Post-procedural rhythm monitoring follows the study protocol.
  Arms: Pulmonary Vein Isolation (PVI) only Group

SUMMARY:
To date, no optimal treatment has been established to improve outcomes in patients with persistent atrial fibrillation. The safety and efficacy of pulsed-field ablation (PFA) have been demonstrated in several studies, and its clinical application is expanding.

- In patients with persistent atrial fibrillation, can the addition of posterior wall isolation (PWI) following pulmonary vein isolation (PVI) using PFA reduce recurrence?

Participants will:

* Undergo either PVI alone or PVI with additional left atrial posterior wall isolation (PWI)
* Visit the clinic to assess for recurrence of atrial tachyarrhythmias

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a major cardiovascular disease with a prevalence of approximately 1.2% in the general population. It accounts for 20-25% of ischemic strokes and is associated with about 30% of heart failure cases. Catheter ablation is an interventional rhythm control strategy that has demonstrated superior outcomes compared to antiarrhythmic drugs (AADs) in patients with drug-refractory AF. For paroxysmal AF, pulmonary vein isolation (PVI) using radiofrequency catheter ablation or cryoballoon ablation has been shown to yield better clinical outcomes than medication alone.

However, in persistent AF, additional ablation strategies beyond PVI have been investigated to improve procedural success rates. While previous studies explored the efficacy of linear ablation and complex fractionated electrogram (CFAE) ablation, recent research suggests that these additional ablation strategies do not significantly improve outcomes in persistent AF. As a result, the optimal catheter ablation strategy for persistent AF remains uncertain.

Nonetheless, some studies have proposed left atrial posterior wall isolation (PWI) as a potential adjunct to reduce AF recurrence in patients with persistent AF. Pulsed-field ablation (PFA) has been recognized in both Europe and the United States for its safety and efficacy, offering a catheter ablation technique that enables a more effective and safer PVI. Additionally, PFA-based posterior wall isolation has been reported to facilitate rapid and safe lesion formation.

Thus, this study aims to prospectively and randomly assign patients undergoing PFA for persistent AF to either:

1. PVI alone or
2. PVI with additional left atrial posterior wall isolation (PWI) By comparing outcomes between these two groups, this study seeks to determine the optimal ablation strategy for patients with persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for catheter ablation according to existing clinical guidelines
* Those without clinically significant structural heart disease (e.g., severe mitral regurgitation)
* Those without contraindications to anticoagulation therapy

Exclusion Criteria:

* Atrial fibrillation associated with severe congenital heart disease or structural heart disease
* Patients with contraindications to general anesthesia or sedation for the procedure
* History of prior cardiac surgery (e.g., Maze procedure, coronary artery bypass grafting)
* History of atrial fibrillation catheter ablation within the past 12 months
* Patients with severe left ventricular dysfunction (left ventricular ejection fraction <30%)
* Patients with active internal bleeding
* Patients with contraindications to anticoagulation therapy and antiarrhythmic drugs
* Valvular atrial fibrillation (e.g., mitral stenosis > grade 2, mechanical valve, prior mitral valve repair)
* Patients with severe comorbid conditions
* Patients with an expected survival of less than one year
* Patients with drug or alcohol addiction
* Pregnant or breastfeeding women
* Any other conditions deemed by the investigator to make the patient unsuitable for study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial tachyarrhythmia | Within one year from the time of enrollment, excluding the first three months after the procedure
  Clinical recurrence rate of atrial fibrillation within one year after the procedure.

SECONDARY OUTCOMES:
Peri-procedural complication | Within one year from the time of enrollment
  Major ; brain hemorrhage, thromboembolism , atrial -esophageal fistula, pericardial effusion, tamponade, irreversible phrenic nerve palsy, bleeding requiring transfusion, Pulmonary Vein Stenosis: Minor ; puncture site bleeding not requiring transfusion , groin hematoma, reversible phrenic nerve palsy
Total procedure time | Periprocedural
  total procedure time
Length of hospital stay | Within one year from the time of enrollment
  Length of hospital stay
patient satisfaction | Within one year from the time of enrollment
  Atrial Fibrillation Effect on Quality-of-Life(AFEQT)
Atrial fibrillation burden | Within one year from the time of enrollment
  Atrial fibrillation burden (%) recorded via holter ECG

CONTACTS AND LOCATIONS:
Locations (1):
- Ewha Womans University Mokdong Hospitoal, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns regarding patient confidentiality and the lack of specific consent for data sharing obtained during the study enrollment process.